CLINICAL TRIAL: NCT06323772
Title: Exploration of New Sensitive Clinical Readouts and Biomarkers That Can Be Used As Clinical Endpoints Tailored to Monitor Treatment Effects in PDE6A-, PDE6B- and RHO-linked Retinitis Pigmentosa: a Non-interventional Trial
Brief Title: Natural History Study in Patients with PDE6A-, PDE6B- and RHO-linked Retinitis Pigmentosa
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: RDC-RP-01
Record Dates: First submitted 2024-03-07; First posted 2024-03-21 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinal Diseases; Eye Diseases; Eye Diseases, Hereditary; Retinal Dystrophies; Retinal Degeneration; Genetic Diseases, Inborn; Retinitis Pigmentosa; PDE6A, PDE6B, RHO; gene therapy trial
MeSH Terms: conditions — Retinitis Pigmentosa; Retinal Diseases; Eye Diseases; Eye Diseases, Hereditary; Retinal Dystrophies; Retinal Degeneration; Genetic Diseases, Inborn; Night Blindness, Congenital Stationary, Autosomal Dominant 2; Night Blindness, Congenital Stationary, Autosomal Dominant 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- PDE6A patients: 15 patients with mutation in PDE6A
- PDE6B patients: 15 patients with mutation in PDE6B
- RHO patients: 10 patients with mutation in RHO

SUMMARY:
The aim of the study is to apply a novel clinical investigation protocol in patients with Phosphodiesterase 6A (PDE6A), PDE6B and Rhodopsin (RHO)-based retinitis pigmentosa. This novel, multimodal clinical examination protocol describes and correlates structural, functional and metabolic aspects during natural disease development.

Test-retest variability of new measurements as well as correlations of the structural, functional, and metabolic changes will be defined to be able to define well-suited readouts for safety and efficacy of future treatment developments before they reach the clinical phase.

DETAILED DESCRIPTION:
Hereditary retinal diseases such as retinitis pigmentosa are rare genetic diagnoses of the retina with chronic lifelong progression, often leading to blindness. Progression varies greatly between individuals. PDE6A, PDE6B and RHO related retinitis pigmentosa phenotypes are typical retinal dystrophies with early onset of rod dysfunctions and a rather slow progression of the cone dysfunction with progression to complete blindness in later adulthood.

Classical gene therapy could improve the function of the rods if successful, although the changes may only be very small and need to be measured using sensitive methods. In contrast, neuroprotective therapeutic approaches could slow down these slow processes even further, which would be extremely difficult to prove as clinical efficacy in a future clinical trial with very individual courses.

In order to have clinical examination methods in the future that can prove the safety and efficacy of neuroprotective approaches, very sensitive examination methods are needed whose test variability is also known. In addition, a neuroprotective treatment method can positively influence the metabolic state of the retina, which, in contrast to slowing down a slow degeneration process, would be a demonstrable effect if the metabolism of the retina can be examined in a clinically relevant way.

For these reasons, the investigators will focus on the above-mentioned genotypes of retinitis pigmentosa in a non-interventional study in order to collect and correlate structural, functional and metabolic examinations of the retina.

ELIGIBILITY:
Inclusion Criteria:

* Age: from 5 years of age
* Patient with PDE6A, PDE6B, and RHO-based retinitis pigmentosa
* Patient and/or legal representatives are willing and able to give written informed consent

Exclusion Criteria:

* severe general disease, that would make longer examinations not possible

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 40 patients with PDE6A, PDE6B, and RHO-based retinitis pigmentosa
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Optical coherence tomography (OCT) | 3-5 years
  OCT volume scans of the macular region, morphological examination
Fundus autofluorescence imaging | 3-5 years
  Fundus autofluorescence imaging, morphological examination
Wide-field fundus photography | 3-5 years
  Wide-field fundus photography, morphological examination
Adaptive optics imaging | 3-5 years
  Adaptive optics imaging, morphological examination
V1 morphology (MRI) | 3-5 years
  MRI, morphological examination
Diffusion Tensor Imaging (DTI) | 3-5 years
  DTI of the optical pathway , morphological examination
flavoprotein fluorescence (FPF) | 3-5 years
  FPF, metabolic readout
Retinal oxymetry | 3-5 years
  Retinal oxymetry, metabolic readout , Local dark adapted adaptation curves
Local dark adapted adaptation curves | 3-5 years
  Local dark adapted adaptation curves , metabolic readout ,
best corrected visual acuity (BCVA) | 3-5 years
  BCVA, functional diagnostics
Static cone perimetry and dark adapted perimetry | 3-5 years
  Static cone perimetry and dark adapted perimetry , functional diagnostics
chromatic pupil campimetry (CPC) | 3-5 years
  scotopic and photopic CPC , functional diagnostics
electroretinogram (ERG) | 3-5 years
  Functional ERG (new flickers 9, 15, 31 Hertz) , functional diagnostics
Virtual reality (VR) functional test | 3-5 years
  VR functional test, functional diagnostics

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Stingl, Prof, Principal Investigator — Department for Opthalmology
Locations (1):
- Institute for Ophthalmic Research, University Tübingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No